CLINICAL TRIAL: NCT04429802
Title: The Effect of Prucalopride (Resolor®) on Gastric Motor Function and Gastric Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: S55741
Record Dates: First submitted 2018-08-24; First posted 2020-06-12 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Gastrointestinal Motility Disorder; Dyspepsia
Keywords: gastric accommodation; gastric sensitivity; gastric compliance; nutrient tolerance
MeSH Terms: conditions — Dyspepsia | interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo is an opaque empty gel capsule obtained from the UZ Gasthuisberg pharmacy. These capsules are composed of 100% gelatine that will rapidly dissolve (disintegration time is 15 minutes) in the stomach without affecting the gastric motor function.
  Interventions: Drug: Placebo
- Prucalopride (Experimental): 2 mg, Resolor®, Shire, Belgium Prucalopride (2 mg) is rapidly absorbed; after a single oral dose of 2 mg Cmax was attained in 2-3 hours. The absolute oral bioavailability is >90%. Concomitant intake of food does not influence the oral bioavailability of prucalopride.
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Drug: Prucalopride — Orally administered
  Other Names: Resolor
  Arms: Prucalopride
Drug: Placebo — Orally administered
  Arms: Placebo

SUMMARY:
Functional Dyspepsia-Postprandial Distress Syndrome (FD-PDS), is characterized by meal-related symptoms such as early satiation and postprandial fullness. Disturbances of gastric motor function have been implicated the pathogenesis of PDS symptoms, and hence, motility modifying agents are considered for the treatment of PDS. Prucalopride (Resolor®), a highly selective 5-TH4 receptor agonist which stimulates gastrointestinal motility throughout the GI tract, is currently approved for the treatment of chronic constipation. The objective of this study was to evaluate the effect of prucalopride on gastric sensorimotor function in healthy volunteers (HV). Methods A total of 17 HV (59% females, mean age 29.4±2.7 years) underwent a barostat and intragastric pressure (IGP) measurements after treatment with placebo or prucalopride (2 mg) in a single blinded cross-over fashion. Isobaric distentions with stepwise increments of 2 mm Hg starting from minimal distending pressure (MDP) and scoring of intensities of gastric sensations (0-6: pain) were used to determine gastric compliance and sensitivity. Gastric accommodation (GA) was quantified as the difference (delta) in intra-balloon volume 30 min before and 60 min after ingestion of 200 ml of a nutrient drink (ND) (1.5 kcal mL(-1)). GA measured by IGP was quantified as the drop of IGP from baseline during the intragastric infusion of ND until maximal satiation. During all tests, epigastric symptoms were scored every 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, male and females, between 18-60 years old

Exclusion Criteria:

Subjects that:

* They are older than 60 years old.
* Have severely decreased kidney function.
* Have severely decreased liver function.
* Have severe heart disease, for example a history of irregular heartbeats, angina or heart attack.
* Have severe lung disease.
* Have severe psychiatric illness or neurological illness.
* Have any gastrointestinal disease
* Women that are pregnant or breastfeeding.
* Have a rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption (Resolor tablets contain lactose).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2016-10-03 (Actual)

PRIMARY OUTCOMES:
The effect of prucalopride on gastric accommodation with gastric barostat technique | 90 minutes
  Gastric barostat: The gastric balloon will be distended at the minimal distending pressure plus 2 mmHg for 90 minutes. During this time, the subject will score their gastric satiation (0-5) every 5 minutes. After the first 30 minutes, the subject will be asked to drink a liquid meal (20 ml Nutridrink, Nutricia; 630 KJ, 6 g proteins, 18.4 g carbohydrates, and 5.8 g lipids per 100 mL) to induce gastric accommodation.
The effect of prucalopride on gastric accommodation with intragastric pressure measurement technique | 60 minutes
  Intragastric pressure measurement with high resolution manometry. A manometry probe, a small, flexible tube, will be passed through the nose into the stomach of the subject. The probe contains 36 channels that measure pressure. The manometry probe will be positioned in the fundus and the position will be then verified by fluoroscopy.
  To infuse the nutrient drink directly into the stomach, a second infusion catheter will be positioned through the mouth of the subject. nutrient drink (Nutridrink, Nutricia) will be infused directly into the stomach at a constant speed of 60 millilitres per minute. Infusion is stopped when the subject reports maximal satiation.

SECONDARY OUTCOMES:
Visual Analog Score for sensitivity | 120 minutes
  Gastric sensitivity will be done by means of step-wise distention of the gastric barostat with Visual Analog Score for sensitivity
The effect of prucalopride on gastric compliance | 120 minutes
  Gastric compliance of the gastric wall will be assessed with step-wise distention of the gastric balloon
The effect of prucalopride on nutrient tolerance | 30 minutes
  The amount of ingested calories will be assessed during intragastric infusion of a nutrient drink will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carbone F, Vanuytsel T, Tack J. The effect of prucalopride on gastric sensorimotor function and satiation in healthy volunteers. Neurogastroenterol Motil. 2021 Aug;33(8):e14083. doi: 10.1111/nmo.14083. Epub 2021 Feb 2. PMID 33615630